CLINICAL TRIAL: NCT04152395
Title: Study of Metabolic Syndrome in Patients Undergoing Endovascular Aortic Repair (EVAR)
Brief Title: Metabolic Syndrome in Patients Undergoing Endovascular Aortic Repair (EVAR)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Elena Arnaoutoglou, Professor of Anesthesiology, University of Thessaly
Other Study IDs: Metabolic syndrome in EVAR
Record Dates: First submitted 2019-09-24; First posted 2019-11-05 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Metabolic Syndrome; Endovascular Aortic Repair
Keywords: Metabolic Syndrome; EVAR
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Metabolic group: Patients with metabolic syndrome undergoing EVAR
  Interventions: Other: EVAR
- Control group: Patients without metabolic syndrome undergoing EVAR
  Interventions: Other: EVAR

INTERVENTIONS:
Other: EVAR — Patients undergoing EVAR

SUMMARY:
This prospective study aims to identify the prevalence of metabolic syndrome in patients undergoing EVAR and the implications of metabolic syndrome on the postoperative outcome, the major complications, the thromboembolic events and the perioperative mortality and morbidity of the patients undergoing vascular surgery.

DETAILED DESCRIPTION:
Patients scheduled for elective EVAR will be randomly divided in two groups. One group patients with metabolic syndrome and one without.

Metabolic syndrome is defined by the definition of 2009 as:

Increased waist circumflex (>94 cm in men and > 80 cm in women), increased triglycerides or in therapy, decreased HDL (< 40 mg/dl in men and <50mg/dl in women) or in therapy, Increased blood pressure (Systolic Blood Pressure>130 mmHg or Diastolic Blood Pressure>85 mmHg) or in therapy, increased fasting glucose (>100mg/dl) or in therapy.

All the patients will be monitored throughout the perioperative period, at 30 days, 6 and 12 months, and any major or minor complication will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* elective EVAR

Exclusion Criteria:

* Patients incapable to give informed consent
* Pregnancy
* Cancer
* Systematic Inflammatory disease
* Use of steroids
* Emergency surgery
* Prior ICU admission

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for elective EVAR
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-12-11 (Estimated); Study Completion 2022-12-11 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 days
  Patients after EVAR who died in 30 days
Mortality | 6 months
  Patients after EVAR who died in 6 months
Mortality | 12 months
  Patients after EVAR who died in 12 months

SECONDARY OUTCOMES:
Systematic inflammatory response | 30 days
  Patients after EVAR that develop Systematic inflammatory response
Systematic inflammatory response | 6 months
  Patients after EVAR that develop Systematic inflammatory response
Systematic inflammatory response | 12 months
  Patients after EVAR that develop Systematic inflammatory response
Postimplantation syndrome | 30 days
  Patients after EVAR that develop Postimplantation syndrome
Postimplantation syndrome | 6 months
  Patients after EVAR that develop Postimplantation syndrome
Postimplantation syndrome | 12 months
  Patients after EVAR that develop Postimplantation syndrome
Renal insufficiency | 30 days
  Patients after EVAR that develop Renal insufficiency
Renal insufficiency | 6 months
  Patients after EVAR that develop Renal insufficiency
Renal insufficiency | 12 months
  Patients after EVAR that develop Renal insufficiency
Cardiovascular events | 30 days
  Incidence of cardiovascular events in patients after EVAR
Cardiovascular events | 6 months
  Incidence of cardiovascular events in patients after EVAR
Cardiovascular events | 12 months
  Incidence of cardiovascular events in patients after EVAR
Thromboembolic events | 30 days
  Incidence of thromboembolic events in patients after EVAR
Thromboembolic events | 6 months
  Incidence of thromboembolic events in patients after EVAR
Thromboembolic events | 12 months
  Incidence of thromboembolic events in patients after EVAR
Complications of surgical procedure | 30 days
  Incidence of Complications of surgical procedure
Complications of surgical procedure | 6 months
  Incidence of Complications of surgical procedure
Complications of surgical procedure | 12 months
  Incidence of Complications of surgical procedure

OTHER OUTCOMES:
Postoperative delirium (POD) | 30 days, 6 and 12 months
  Prevalence of POD in patients undergoing EVAR

CONTACTS AND LOCATIONS:
Overall Officials: Elena Arnaoutoglou, MD, PhD, Study Chair — University of Thessaly; Haralampos Milionis, MD, PhD, Study Director — University of Ioannina; Konstantina Kolonia, MD, PhD, Principal Investigator — University Hospital of Larissa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Alberti KG, Eckel RH, Grundy SM, Zimmet PZ, Cleeman JI, Donato KA, Fruchart JC, James WP, Loria CM, Smith SC Jr; International Diabetes Federation Task Force on Epidemiology and Prevention; Hational Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; International Association for the Study of Obesity. Harmonizing the metabolic syndrome: a joint interim statement of the International Diabetes Federation Task Force on Epidemiology and Prevention; National Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; and International Association for the Study of Obesity. Circulation. 2009 Oct 20;120(16):1640-5. doi: 10.1161/CIRCULATIONAHA.109.192644. Epub 2009 Oct 5. PMID 19805654
- [Result] Alberti KG, Zimmet P, Shaw J; IDF Epidemiology Task Force Consensus Group. The metabolic syndrome--a new worldwide definition. Lancet. 2005 Sep 24-30;366(9491):1059-62. doi: 10.1016/S0140-6736(05)67402-8. No abstract available. PMID 16182882
- [Result] Grundy SM, Cleeman JI, Daniels SR, Donato KA, Eckel RH, Franklin BA, Gordon DJ, Krauss RM, Savage PJ, Smith SC Jr, Spertus JA, Fernando Costa. Diagnosis and management of the metabolic syndrome: an American Heart Association/National Heart, Lung, and Blood Institute scientific statement: Executive Summary. Crit Pathw Cardiol. 2005 Dec;4(4):198-203. doi: 10.1097/00132577-200512000-00018. No abstract available. PMID 18340209
- [Result] Aguilar M, Bhuket T, Torres S, Liu B, Wong RJ. Prevalence of the metabolic syndrome in the United States, 2003-2012. JAMA. 2015 May 19;313(19):1973-4. doi: 10.1001/jama.2015.4260. No abstract available. PMID 25988468